CLINICAL TRIAL: NCT01515124
Title: The Women In Steady Exercise Research (WISER) Survivor Trial & Cost of Illness and Cost Effectiveness of Alternative Management Strategies
Brief Title: The Women In Steady Exercise Research (WISER) Survivor Trial
Acronym: WISER Survivor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: U54CA155850 (NIH)
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Lymphedema
Keywords: Lymphedema; Strength training intervention; Weight loss intervention; Breast cancer recurrence; Cost Effectiveness
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All participants asked at the start of each measurement encounter not to inform measurement staff of their randomization group status. All measurement staff asked to guess group status at end of each measurement encounter. Patterns of responses beyond chance result in corrective action to improve masking (e.g.; requests from PI for participants to mask group status)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lymphedema Care Only (No Intervention): All 4 groups receive lymphedema care as follows:
  1. 2 custom fitted compression garments (baseline and 6 months)
  2. evaluations for flare-ups at request (and at each measurement time point)
  3. lymphedema treatment by a certified lymphatic therapist upon detection of a flare-up, paid for by the study. No limit was placed on number of sessions.
- Exercise only (Experimental): The Exercise Intervention combines 60-90 minute twice-weekly supervised weight-lifting sessions with 180 minutes of weekly aerobic exercise. Women will be trained by certified fitness professionals in both the weight-lifting intervention and in safely increasing their aerobic exercise activity over 6 weekly sessions, and then monitored through phone contact, and monthly in-person sessions. All exercise participants will be provided with 'Power Blocks' which are adjustable dumbbells with which they can increase resistance in 1-2 pound increments from 1-21 pounds. All weight training will be done in their homes except for the first 6 weekly session and monthly check-in sessions. Exercise only group members also received the Lymphedema care intervention described above.
  Interventions: Behavioral: Exercise Intervention
- Weight loss only (Experimental): The Weight Loss Intervention begins with a 24 week intensive phase that includes weekly meetings and provision of all meals and snacks from a commercial manufacturer (NutriSystem®, Inc., Fort Washington, PA). Daily caloric intake will be strictly controlled during this first 24 weeks at 1200-1500 calories per day. Participants will be guided to stay at the same number of calories per day until reaching goal weight, followed by a gradual increase in caloric intake (of approximately 500 calories/d) to maintain their weight throughout the remainder of the intervention. The treatment groups will be led by registered dietitians and will receive ongoing supervision via telephone and email contact. Weight loss only group members also received the Lymphedema care intervention described above.
  Interventions: Behavioral: Weight Loss Intervention
- Exercise and Weight loss combined (Experimental): Participants in this group will receive a combination of the supervised twice-weekly weight training sessions and the weight loss program. Combined group members also received the Lymphedema care intervention described above.
  Interventions: Behavioral: Exercise Intervention; Behavioral: Weight Loss Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — The Exercise Intervention combines the twice-weekly weight-lifting intervention from PAL with the 180 minutes of weekly aerobic exercise from the recently completed WISER trial and the ongoing WISER Sister Trial. Women will be trained by certified fitness professionals in both the PAL weight-lifting intervention and in safely increasing their aerobic exercise activity over 6 weekly sessions, and then monitored through phone contact, and monthly in-person sessions.
  Arms: Exercise and Weight loss combined; Exercise only
Behavioral: Weight Loss Intervention — The Weight Loss Intervention begins with a 24 week intensive phase that includes weekly meetings and provision of all meals and snacks from a commercial manufacturer (NutriSystem, Inc., Fort Washington, PA). Daily caloric intake will be strictly controlled during this first 24 weeks at 1200-1500 calories per day.
  Arms: Exercise and Weight loss combined; Weight loss only

SUMMARY:
WISER Survivor is a one year weight loss and exercise study for sedentary breast cancer survivors who are overweight or obese with breast cancer related lymphedema. There will be four groups in this trial: exercise only, weight loss only, exercise and weight-loss combined, and a control group. The primary purpose of this study is to test the effects of these interventions on clinical lymphedema outcomes. Secondary outcomes include weight loss, breast cancer related biomarkers, and quality of life. To the extent that funding will be available, participants will be followed long term to examine effects on recurrence and mortality.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer survivor
* overweight or obese (BMI of 25 or greater)
* must have breast cancer related lymphedema
* at least 6 months post-treatment (e.g. surgery, chemotherapy, or radiotherapy) but there will be no upper limit on time elapsed from diagnosis
* the eligible age range will have no lower limit.
* currently free of cancer

Exclusion Criteria:

* medical conditions or medications that would prohibit participation in an exercise program or would negatively impact our ability to test our primary aims
* inability to walk for 6 minutes unaided
* extremely obese (body mass index greater or equal to 50 kg/m2)
* plans for additional (e.g. curative or reconstructive) surgery during the study period
* self-report of weight-lifting within the past year
* already engaging in 3 or more times weekly aerobic activity of moderate intensity
* planning to move away from the area over the next year
* current use of weight loss medication (OTC or prescription)
* self-report of alcohol or substance abuse within the past 12 months, including at-risk drinking (current consumption of more than 14 alcoholic drinks per week)
* weight loss of greater than 10 % in the past 3 months
* history of bariatric surgery
* women who are pregnant

Max Age: 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Percent interlimb difference, change over 12 months. | Baseline and 12 months
  Arm volumes for affected and unaffected limbs will be measured by perometry and the % difference will be determined at baseline and 12 months. the absolute percentage point difference of differences (% interlimb difference at 12 months minus % interlimb difference at baseline) will be the primary outcome

SECONDARY OUTCOMES:
Clinical Lymphedema Events | Data collected over the 12 month follow-up, with events collected as reported
  Flare-ups and cellulitic infections (number and type recorded)
Clinical Evaluation Score for Lymphedema | Baseline and 12 months
  Standardized clinical evaluation survey completed by certified lymphatic therapists
Norman Lymphedema Survey | Baseline and 12 months
  Thirteen symptoms, recorded within a standardized survey (Norman Lymphedema Survey)
Weight loss | Baseline and 12 months
  body weight loss over 12 months
Biomarkers: Estradiol | baseline and 12 months
  circulating estradiol levels in the blood
Biomarkers: Testosterone | baseline and 12 months
  circulating testosterone levels in the blood
Biomarkers - Sex Hormone Binding Globulin | baseline and 12 months
  circulating sex hormone binding globulin levels in the blood
Inflammation: Interleukin six | baseline and 12 months
  Circulating interleukin six levels in the blood
Inflammation: C reactive protein | baseline and 12 months
  Circulating c reactive protein levels in the blood
Adiponectin | baseline and 12 months
  circulating Adiponectin levels in the blood
Leptin | baseline and 12 months
  circulating leptin levels in the blood
F2-isoprostanes | baseline and 12 months
  circulating F2-isoprostane levels in the blood
Insulin | baseline and 12 months
  circulating insulin levels in the blood
Glucose | baseline and 12 months
  circulating glucose levels in the blood
insulin like growth factor one | baseline and 12 months
  circulating levels of insulin like growth factor one in the blood
insulin like growth factor binding protein three | baseline and 12 months
  circulating levels of insulin like growth factor binding protein three in the blood
Upper limb lymphedema twenty seven | baseline and 12 months
  27 item survey on lymphedema quality of life
body image and relationship survey | baseline and 12 months
  32 item survey on body image specifically developed for breast cancer survivors

OTHER OUTCOMES:
breast cancer recurrence | 10 years post trial
  participants will be followed for breast cancer recurrence
mortality | 10 years post trial
  participants will be followed for mortality

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn H. Schmitz, MPH,PhD, Principal Investigator — Penn State University
Locations (1):
- The Penn TREC Survivorship Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Speck RM, Courneya KS, Masse LC, Duval S, Schmitz KH. An update of controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. J Cancer Surviv. 2010 Jun;4(2):87-100. doi: 10.1007/s11764-009-0110-5. Epub 2010 Jan 6. PMID 20052559
- [Background] Hewitt M, Greenfield, S., Stovall, E. , ed. From Cancer Patient to Cancer Survivor: Lost in Transition. Washington, D.C.: National Academies Press; 2006.
- [Background] Smith BD, Smith GL, Hurria A, Hortobagyi GN, Buchholz TA. Future of cancer incidence in the United States: burdens upon an aging, changing nation. J Clin Oncol. 2009 Jun 10;27(17):2758-65. doi: 10.1200/JCO.2008.20.8983. Epub 2009 Apr 29. PMID 19403886
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Hursting SD, Lashinger LM, Colbert LH, Rogers CJ, Wheatley KW, Nunez NP, Mahabir S, Barrett JC, Forman MR, Perkins SN. Energy balance and carcinogenesis: underlying pathways and targets for intervention. Curr Cancer Drug Targets. 2007 Aug;7(5):484-91. doi: 10.2174/156800907781386623. PMID 17691908
- [Background] Holmes MD, Chen WY, Feskanich D, Kroenke CH, Colditz GA. Physical activity and survival after breast cancer diagnosis. JAMA. 2005 May 25;293(20):2479-86. doi: 10.1001/jama.293.20.2479. PMID 15914748
- [Background] Friedenreich CM, Gregory J, Kopciuk KA, Mackey JR, Courneya KS. Prospective cohort study of lifetime physical activity and breast cancer survival. Int J Cancer. 2009 Apr 15;124(8):1954-62. doi: 10.1002/ijc.24155. PMID 19123472
- [Background] Irwin ML, Smith AW, McTiernan A, Ballard-Barbash R, Cronin K, Gilliland FD, Baumgartner RN, Baumgartner KB, Bernstein L. Influence of pre- and postdiagnosis physical activity on mortality in breast cancer survivors: the health, eating, activity, and lifestyle study. J Clin Oncol. 2008 Aug 20;26(24):3958-64. doi: 10.1200/JCO.2007.15.9822. PMID 18711185
- [Background] Armer JM. The problem of post-breast cancer lymphedema: impact and measurement issues. Cancer Invest. 2005;23(1):76-83. PMID 15779870
- [Background] Norman SA, Localio AR, Potashnik SL, Simoes Torpey HA, Kallan MJ, Weber AL, Miller LT, Demichele A, Solin LJ. Lymphedema in breast cancer survivors: incidence, degree, time course, treatment, and symptoms. J Clin Oncol. 2009 Jan 20;27(3):390-7. doi: 10.1200/JCO.2008.17.9291. Epub 2008 Dec 8. PMID 19064976
- [Background] Francis WP, Abghari P, Du W, Rymal C, Suna M, Kosir MA. Improving surgical outcomes: standardizing the reporting of incidence and severity of acute lymphedema after sentinel lymph node biopsy and axillary lymph node dissection. Am J Surg. 2006 Nov;192(5):636-9. doi: 10.1016/j.amjsurg.2006.08.018. No abstract available. PMID 17071198
- [Background] Schrenk P, Rieger R, Shamiyeh A, Wayand W. Morbidity following sentinel lymph node biopsy versus axillary lymph node dissection for patients with breast carcinoma. Cancer. 2000 Feb 1;88(3):608-14. doi: 10.1002/(sici)1097-0142(20000201)88:33.0.co;2-k. PMID 10649254
- [Background] Wilke LG, McCall LM, Posther KE, Whitworth PW, Reintgen DS, Leitch AM, Gabram SG, Lucci A, Cox CE, Hunt KK, Herndon JE 2nd, Giuliano AE. Surgical complications associated with sentinel lymph node biopsy: results from a prospective international cooperative group trial. Ann Surg Oncol. 2006 Apr;13(4):491-500. doi: 10.1245/ASO.2006.05.013. Epub 2006 Mar 2. PMID 16514477
- [Background] Petrek JA, Heelan MC. Incidence of breast carcinoma-related lymphedema. Cancer. 1998 Dec 15;83(12 Suppl American):2776-81. doi: 10.1002/(sici)1097-0142(19981215)83:12b+3.0.co;2-v. PMID 9874397
- [Background] Shih YC, Xu Y, Cormier JN, Giordano S, Ridner SH, Buchholz TA, Perkins GH, Elting LS. Incidence, treatment costs, and complications of lymphedema after breast cancer among women of working age: a 2-year follow-up study. J Clin Oncol. 2009 Apr 20;27(12):2007-14. doi: 10.1200/JCO.2008.18.3517. Epub 2009 Mar 16. PMID 19289624
- [Background] Maunsell E, Brisson J, Deschenes L. Psychological distress after initial treatment for breast cancer: a comparison of partial and total mastectomy. J Clin Epidemiol. 1989;42(8):765-71. doi: 10.1016/0895-4356(89)90074-7. PMID 2760668
- [Background] Passik SD, McDonald MV. Psychosocial aspects of upper extremity lymphedema in women treated for breast carcinoma. Cancer. 1998 Dec 15;83(12 Suppl American):2817-20. doi: 10.1002/(sici)1097-0142(19981215)83:12b+3.0.co;2-2. PMID 9874404
- [Background] Sneeuw KC, Aaronson NK, Yarnold JR, Broderick M, Regan J, Ross G, Goddard A. Cosmetic and functional outcomes of breast conserving treatment for early stage breast cancer. 2. Relationship with psychosocial functioning. Radiother Oncol. 1992 Nov;25(3):160-6. doi: 10.1016/0167-8140(92)90262-s. PMID 1470692
- [Background] Carter BJ. Women's experiences of lymphedema. Oncol Nurs Forum. 1997 Jun;24(5):875-82. PMID 9201739
- [Background] Ahmed RL, Prizment A, Lazovich D, Schmitz KH, Folsom AR. Lymphedema and quality of life in breast cancer survivors: the Iowa Women's Health Study. J Clin Oncol. 2008 Dec 10;26(35):5689-96. doi: 10.1200/JCO.2008.16.4731. Epub 2008 Nov 10. PMID 19001331
- [Background] McWayne J, Heiney SP. Psychologic and social sequelae of secondary lymphedema: a review. Cancer. 2005 Aug 1;104(3):457-66. doi: 10.1002/cncr.21195. PMID 15968692
- [Background] Cheville A. Patient perceptions of lymphedema maintenance therapy: is the cure worse than the condition? In: American Academy of Physical Medicine and Rehabilitation Orlando, FL; 2002.
- [Background] Mak SS, Yeo W, Lee YM, Tse SM, Ho FP, Zee B, Chan E. Risk factors for the initiation and aggravation of lymphoedema after axillary lymph node dissection for breast cancer. Hong Kong Med J. 2009 Jun;15(3 Suppl 4):8-12. No abstract available. PMID 19509430
- [Background] Bar Ad V, Cheville A, Solin LJ, Dutta P, Both S, Harris EE. Time course of mild arm lymphedema after breast conservation treatment for early-stage breast cancer. Int J Radiat Oncol Biol Phys. 2010 Jan 1;76(1):85-90. doi: 10.1016/j.ijrobp.2009.01.024. PMID 19427748
- [Background] Cheville AL, Almoza M, Courmier JN, Basford JR. A prospective cohort study defining utilities using time trade-offs and the Euroqol-5D to assess the impact of cancer-related lymphedema. Cancer. 2010 Aug 1;116(15):3722-31. doi: 10.1002/cncr.25068. PMID 20564063
- [Background] Ridner SH. Quality of life and a symptom cluster associated with breast cancer treatment-related lymphedema. Support Care Cancer. 2005 Nov;13(11):904-11. doi: 10.1007/s00520-005-0810-y. Epub 2005 Apr 6. PMID 15812652
- [Background] Lawenda BD, Mondry TE, Johnstone PA. Lymphedema: a primer on the identification and management of a chronic condition in oncologic treatment. CA Cancer J Clin. 2009 Jan-Feb;59(1):8-24. doi: 10.3322/caac.20001. PMID 19147865
- [Background] Karppelin M, Siljander T, Vuopio-Varkila J, Kere J, Huhtala H, Vuento R, Jussila T, Syrjanen J. Factors predisposing to acute and recurrent bacterial non-necrotizing cellulitis in hospitalized patients: a prospective case-control study. Clin Microbiol Infect. 2010 Jun;16(6):729-34. doi: 10.1111/j.1469-0691.2009.02906.x. Epub 2009 Aug 20. PMID 19694769
- [Background] Schmitz KH. Balancing lymphedema risk: exercise versus deconditioning for breast cancer survivors. Exerc Sport Sci Rev. 2010 Jan;38(1):17-24. doi: 10.1097/JES.0b013e3181c5cd5a. PMID 20016295
- [Background] Cheema B, Gaul CA, Lane K, Fiatarone Singh MA. Progressive resistance training in breast cancer: a systematic review of clinical trials. Breast Cancer Res Treat. 2008 May;109(1):9-26. doi: 10.1007/s10549-007-9638-0. Epub 2007 Jul 12. PMID 17624588
- [Background] Schmitz KH, Ahmed RL, Troxel A, Cheville A, Smith R, Lewis-Grant L, Bryan CJ, Williams-Smith CT, Greene QP. Weight lifting in women with breast-cancer-related lymphedema. N Engl J Med. 2009 Aug 13;361(7):664-73. doi: 10.1056/NEJMoa0810118. PMID 19675330
- [Background] Eder K, Baffy N, Falus A, Fulop AK. The major inflammatory mediator interleukin-6 and obesity. Inflamm Res. 2009 Nov;58(11):727-36. doi: 10.1007/s00011-009-0060-4. Epub 2009 Jun 19. PMID 19543691
- [Background] Shaw C, Mortimer P, Judd PA. A randomized controlled trial of weight reduction as a treatment for breast cancer-related lymphedema. Cancer. 2007 Oct 15;110(8):1868-74. doi: 10.1002/cncr.22994. PMID 17823909
- [Background] Shaw C, Mortimer P, Judd PA. Randomized controlled trial comparing a low-fat diet with a weight-reduction diet in breast cancer-related lymphedema. Cancer. 2007 May 15;109(10):1949-56. doi: 10.1002/cncr.22638. PMID 17393377
- [Background] Schmitz KH, Ahmed RL, Hannan PJ, Yee D. Safety and efficacy of weight training in recent breast cancer survivors to alter body composition, insulin, and insulin-like growth factor axis proteins. Cancer Epidemiol Biomarkers Prev. 2005 Jul;14(7):1672-80. doi: 10.1158/1055-9965.EPI-04-0736. PMID 16030100
- [Background] Holick CN, Newcomb PA, Trentham-Dietz A, Titus-Ernstoff L, Bersch AJ, Stampfer MJ, Baron JA, Egan KM, Willett WC. Physical activity and survival after diagnosis of invasive breast cancer. Cancer Epidemiol Biomarkers Prev. 2008 Feb;17(2):379-86. doi: 10.1158/1055-9965.EPI-07-0771. Epub 2008 Feb 4. PMID 18250341
- [Background] Pierce JP, Stefanick ML, Flatt SW, Natarajan L, Sternfeld B, Madlensky L, Al-Delaimy WK, Thomson CA, Kealey S, Hajek R, Parker BA, Newman VA, Caan B, Rock CL. Greater survival after breast cancer in physically active women with high vegetable-fruit intake regardless of obesity. J Clin Oncol. 2007 Jun 10;25(17):2345-51. doi: 10.1200/JCO.2006.08.6819. PMID 17557947
- [Background] Kroenke CH, Chen WY, Rosner B, Holmes MD. Weight, weight gain, and survival after breast cancer diagnosis. J Clin Oncol. 2005 Mar 1;23(7):1370-8. doi: 10.1200/JCO.2005.01.079. Epub 2005 Jan 31. PMID 15684320
- [Background] Caan BJ, Emond JA, Natarajan L, Castillo A, Gunderson EP, Habel L, Jones L, Newman VA, Rock CL, Slattery ML, Stefanick ML, Sternfeld B, Thomson CA, Pierce JP. Post-diagnosis weight gain and breast cancer recurrence in women with early stage breast cancer. Breast Cancer Res Treat. 2006 Sep;99(1):47-57. doi: 10.1007/s10549-006-9179-y. Epub 2006 Mar 16. PMID 16541317
- [Background] Daniell HW. Weight loss after breast cancer diagnosis may not improve prognosis. J Clin Oncol. 2009 Feb 10;27(5):829-30; author reply 830-1. doi: 10.1200/JCO.2008.20.5294. Epub 2009 Jan 12. No abstract available. PMID 19139422
- [Background] Chlebowski RT, Blackburn GL, Thomson CA, Nixon DW, Shapiro A, Hoy MK, Goodman MT, Giuliano AE, Karanja N, McAndrew P, Hudis C, Butler J, Merkel D, Kristal A, Caan B, Michaelson R, Vinciguerra V, Del Prete S, Winkler M, Hall R, Simon M, Winters BL, Elashoff RM. Dietary fat reduction and breast cancer outcome: interim efficacy results from the Women's Intervention Nutrition Study. J Natl Cancer Inst. 2006 Dec 20;98(24):1767-76. doi: 10.1093/jnci/djj494. PMID 17179478
- [Background] Pierce JP, Natarajan L, Caan BJ, Parker BA, Greenberg ER, Flatt SW, Rock CL, Kealey S, Al-Delaimy WK, Bardwell WA, Carlson RW, Emond JA, Faerber S, Gold EB, Hajek RA, Hollenbach K, Jones LA, Karanja N, Madlensky L, Marshall J, Newman VA, Ritenbaugh C, Thomson CA, Wasserman L, Stefanick ML. Influence of a diet very high in vegetables, fruit, and fiber and low in fat on prognosis following treatment for breast cancer: the Women's Healthy Eating and Living (WHEL) randomized trial. JAMA. 2007 Jul 18;298(3):289-98. doi: 10.1001/jama.298.3.289. PMID 17635889
- [Background] Irwin ML, Varma K, Alvarez-Reeves M, Cadmus L, Wiley A, Chung GG, Dipietro L, Mayne ST, Yu H. Randomized controlled trial of aerobic exercise on insulin and insulin-like growth factors in breast cancer survivors: the Yale Exercise and Survivorship study. Cancer Epidemiol Biomarkers Prev. 2009 Jan;18(1):306-13. doi: 10.1158/1055-9965.EPI-08-0531. PMID 19124513
- [Background] Ligibel JA, Campbell N, Partridge A, Chen WY, Salinardi T, Chen H, Adloff K, Keshaviah A, Winer EP. Impact of a mixed strength and endurance exercise intervention on insulin levels in breast cancer survivors. J Clin Oncol. 2008 Feb 20;26(6):907-12. doi: 10.1200/JCO.2007.12.7357. PMID 18281663
- [Background] Fairey AS, Courneya KS, Field CJ, Bell GJ, Jones LW, Mackey JR. Effects of exercise training on fasting insulin, insulin resistance, insulin-like growth factors, and insulin-like growth factor binding proteins in postmenopausal breast cancer survivors: a randomized controlled trial. Cancer Epidemiol Biomarkers Prev. 2003 Aug;12(8):721-7. PMID 12917202
- [Background] Fairey AS, Courneya KS, Field CJ, Bell GJ, Jones LW, Mackey JR. Randomized controlled trial of exercise and blood immune function in postmenopausal breast cancer survivors. J Appl Physiol (1985). 2005 Apr;98(4):1534-40. doi: 10.1152/japplphysiol.00566.2004. PMID 15772062
- [Background] Fairey AS, Courneya KS, Field CJ, Bell GJ, Jones LW, Martin BS, Mackey JR. Effect of exercise training on C-reactive protein in postmenopausal breast cancer survivors: a randomized controlled trial. Brain Behav Immun. 2005 Sep;19(5):381-8. doi: 10.1016/j.bbi.2005.04.001. PMID 15922556
- [Background] Naumov GN, Folkman J, Straume O. Tumor dormancy due to failure of angiogenesis: role of the microenvironment. Clin Exp Metastasis. 2009;26(1):51-60. doi: 10.1007/s10585-008-9176-0. Epub 2008 Jun 18. PMID 18563595
- [Background] Rock CL, Flatt SW, Laughlin GA, Gold EB, Thomson CA, Natarajan L, Jones LA, Caan BJ, Stefanick ML, Hajek RA, Al-Delaimy WK, Stanczyk FZ, Pierce JP; Women's Healthy Eating and Living Study Group. Reproductive steroid hormones and recurrence-free survival in women with a history of breast cancer. Cancer Epidemiol Biomarkers Prev. 2008 Mar;17(3):614-20. doi: 10.1158/1055-9965.EPI-07-0761. Epub 2008 Mar 6. PMID 18323413
- [Background] Pierce BL, Ballard-Barbash R, Bernstein L, Baumgartner RN, Neuhouser ML, Wener MH, Baumgartner KB, Gilliland FD, Sorensen BE, McTiernan A, Ulrich CM. Elevated biomarkers of inflammation are associated with reduced survival among breast cancer patients. J Clin Oncol. 2009 Jul 20;27(21):3437-44. doi: 10.1200/JCO.2008.18.9068. Epub 2009 May 26. PMID 19470939
- [Background] Ozet A, Arpaci F, Yilmaz MI, Ayta H, Ozturk B, Komurcu S, Yavuz AA, Tezcan Y, Acikel C. Effects of tamoxifen on the serum leptin level in patients with breast cancer. Jpn J Clin Oncol. 2001 Sep;31(9):424-7. doi: 10.1093/jjco/hye097. PMID 11689595
- [Background] Hou WK, Xu YX, Yu T, Zhang L, Zhang WW, Fu CL, Sun Y, Wu Q, Chen L. Adipocytokines and breast cancer risk. Chin Med J (Engl). 2007 Sep 20;120(18):1592-6. PMID 17908478
- [Background] Dai Q, Gao YT, Shu XO, Yang G, Milne G, Cai Q, Wen W, Rothman N, Cai H, Li H, Xiang Y, Chow WH, Zheng W. Oxidative stress, obesity, and breast cancer risk: results from the Shanghai Women's Health Study. J Clin Oncol. 2009 May 20;27(15):2482-8. doi: 10.1200/JCO.2008.19.7970. Epub 2009 Apr 20. PMID 19380446
- [Background] Pasanisi P, Venturelli E, Morelli D, Fontana L, Secreto G, Berrino F. Serum insulin-like growth factor-I and platelet-derived growth factor as biomarkers of breast cancer prognosis. Cancer Epidemiol Biomarkers Prev. 2008 Jul;17(7):1719-22. doi: 10.1158/1055-9965.EPI-07-0654. PMID 18628423
- [Background] Lukanova A, Lundin E, Zeleniuch-Jacquotte A, Muti P, Mure A, Rinaldi S, Dossus L, Micheli A, Arslan A, Lenner P, Shore RE, Krogh V, Koenig KL, Riboli E, Berrino F, Hallmans G, Stattin P, Toniolo P, Kaaks R. Body mass index, circulating levels of sex-steroid hormones, IGF-I and IGF-binding protein-3: a cross-sectional study in healthy women. Eur J Endocrinol. 2004 Feb;150(2):161-71. doi: 10.1530/eje.0.1500161. PMID 14763914
- [Background] Pierce BL, Neuhouser ML, Wener MH, Bernstein L, Baumgartner RN, Ballard-Barbash R, Gilliland FD, Baumgartner KB, Sorensen B, McTiernan A, Ulrich CM. Correlates of circulating C-reactive protein and serum amyloid A concentrations in breast cancer survivors. Breast Cancer Res Treat. 2009 Mar;114(1):155-67. doi: 10.1007/s10549-008-9985-5. Epub 2008 Apr 10. PMID 18401703
- [Background] You T, Berman DM, Ryan AS, Nicklas BJ. Effects of hypocaloric diet and exercise training on inflammation and adipocyte lipolysis in obese postmenopausal women. J Clin Endocrinol Metab. 2004 Apr;89(4):1739-46. doi: 10.1210/jc.2003-031310. PMID 15070939
- [Background] Thomson CA, Giuliano AR, Shaw JW, Rock CL, Ritenbaugh CK, Hakim IA, Hollenbach KA, Alberts DS, Pierce JP. Diet and biomarkers of oxidative damage in women previously treated for breast cancer. Nutr Cancer. 2005;51(2):146-54. doi: 10.1207/s15327914nc5102_4. PMID 15860436
- [Background] Gram IT, Norat T, Rinaldi S, Dossus L, Lukanova A, Tehard B, Clavel-Chapelon F, van Gils CH, van Noord PA, Peeters PH, Bueno-de-Mesquita HB, Nagel G, Linseisen J, Lahmann PH, Boeing H, Palli D, Sacerdote C, Panico S, Tumino R, Sieri S, Dorronsoro M, Quiros JR, Navarro CA, Barricarte A, Tormo MJ, Gonzalez CA, Overvad K, Paaske Johnsen S, Olsen A, Tjonneland A, Travis R, Allen N, Bingham S, Khaw KT, Stattin P, Trichopoulou A, Kalapothaki V, Psaltopoulou T, Casagrande C, Riboli E, Kaaks R. Body mass index, waist circumference and waist-hip ratio and serum levels of IGF-I and IGFBP-3 in European women. Int J Obes (Lond). 2006 Nov;30(11):1623-31. doi: 10.1038/sj.ijo.0803324. Epub 2006 Mar 21. PMID 16552400
- [Background] Seaman S, Stevens J, Yang MY, Logsdon D, Graff-Cherry C, St Croix B. Genes that distinguish physiological and pathological angiogenesis. Cancer Cell. 2007 Jun;11(6):539-54. doi: 10.1016/j.ccr.2007.04.017. PMID 17560335
- [Background] Vona-Davis L, Rose DP. Angiogenesis, adipokines and breast cancer. Cytokine Growth Factor Rev. 2009 Jun;20(3):193-201. doi: 10.1016/j.cytogfr.2009.05.007. Epub 2009 Jun 10. PMID 19520599
- [Background] Hieken TJ, Cheregi J, Farolan M, Kim J, Velasco JM. Predicting relapse in ductal carcinoma in situ patients: an analysis of biologic markers with long-term follow-up. Am J Surg. 2007 Oct;194(4):504-6. doi: 10.1016/j.amjsurg.2007.07.002. PMID 17826066
- [Background] Nicolini A, Campani D, Miccoli P, Spinelli C, Carpi A, Menicagli M, Ferrari P, Gadducci G, Rossi G, Fini M, Giavaresi G, Bonazzi V, Giardino R. Vascular endothelial growth factor (VEGF) and other common tissue prognostic indicators in breast cancer: a case-control study. Int J Biol Markers. 2004 Oct-Dec;19(4):275-81. doi: 10.1177/172460080401900404. PMID 15646833
- [Background] Linderholm BK, Hellborg H, Johansson U, Elmberger G, Skoog L, Lehtio J, Lewensohn R. Significantly higher levels of vascular endothelial growth factor (VEGF) and shorter survival times for patients with primary operable triple-negative breast cancer. Ann Oncol. 2009 Oct;20(10):1639-46. doi: 10.1093/annonc/mdp062. Epub 2009 Jun 23. PMID 19549711
- [Background] Shivakumar S, Prabhakar BT, Jayashree K, Rajan MG, Salimath BP. Evaluation of serum vascular endothelial growth factor (VEGF) and microvessel density (MVD) as prognostic indicators in carcinoma breast. J Cancer Res Clin Oncol. 2009 Apr;135(4):627-36. doi: 10.1007/s00432-008-0497-9. Epub 2008 Oct 21. PMID 18936974
- [Background] Calleri A, Bono A, Bagnardi V, Quarna J, Mancuso P, Rabascio C, Dellapasqua S, Campagnoli E, Shaked Y, Goldhirsch A, Colleoni M, Bertolini F. Predictive Potential of Angiogenic Growth Factors and Circulating Endothelial Cells in Breast Cancer Patients Receiving Metronomic Chemotherapy Plus Bevacizumab. Clin Cancer Res. 2009 Dec 15;15(24):7652-7657. doi: 10.1158/1078-0432.CCR-09-1493. PMID 19996223
- [Background] Zaslavsky A, Baek KH, Lynch RC, Short S, Grillo J, Folkman J, Italiano JE Jr, Ryeom S. Platelet-derived thrombospondin-1 is a critical negative regulator and potential biomarker of angiogenesis. Blood. 2010 Jun 3;115(22):4605-13. doi: 10.1182/blood-2009-09-242065. Epub 2010 Jan 19. PMID 20086246
- [Background] Speck RM, Gross CR, Hormes JM, Ahmed RL, Lytle LA, Hwang WT, Schmitz KH. Changes in the Body Image and Relationship Scale following a one-year strength training trial for breast cancer survivors with or at risk for lymphedema. Breast Cancer Res Treat. 2010 Jun;121(2):421-30. doi: 10.1007/s10549-009-0550-7. Epub 2009 Sep 22. PMID 19771507
- [Background] Hormes JM, Bryan C, Lytle LA, Gross CR, Ahmed RL, Troxel AB, Schmitz KH. Impact of lymphedema and arm symptoms on quality of life in breast cancer survivors. Lymphology. 2010 Mar;43(1):1-13. PMID 20552814
- [Background] Weiss JM, Spray BJ. The effect of complete decongestive therapy on the quality of life of patients with peripheral lymphedema. Lymphology. 2002 Jun;35(2):46-58. PMID 12081052
- [Background] Carver JR, Shapiro CL, Ng A, Jacobs L, Schwartz C, Virgo KS, Hagerty KL, Somerfield MR, Vaughn DJ; ASCO Cancer Survivorship Expert Panel. American Society of Clinical Oncology clinical evidence review on the ongoing care of adult cancer survivors: cardiac and pulmonary late effects. J Clin Oncol. 2007 Sep 1;25(25):3991-4008. doi: 10.1200/JCO.2007.10.9777. Epub 2007 Jun 18. PMID 17577017
- [Background] Schmitz KH, Troxel AB, Cheville A, Grant LL, Bryan CJ, Gross CR, Lytle LA, Ahmed RL. Physical Activity and Lymphedema (the PAL trial): assessing the safety of progressive strength training in breast cancer survivors. Contemp Clin Trials. 2009 May;30(3):233-45. doi: 10.1016/j.cct.2009.01.001. Epub 2009 Jan 8. PMID 19171204
- [Background] Ohira T, Schmitz KH, Ahmed RL, Yee D. Effects of weight training on quality of life in recent breast cancer survivors: the Weight Training for Breast Cancer Survivors (WTBS) study. Cancer. 2006 May 1;106(9):2076-83. doi: 10.1002/cncr.21829. PMID 16568409
- [Background] Derbas J, Vetter, M., Volger, S., Khan, Z., Panigrahi, E., Tsai, A.G., Sarwer, D.B., Wadden, T.A. Improving Weight Management in Primary Care Practice: A Possible Role for Auxiliary Health Professionals Collaborating with Primary Care Physicians. Obesity and Weight Management 2009;5:210-5.
- [Background] Klemp JK CS, Papsek S, et al. . Feasibility of a diet, exercise, and behavior modification intervention for post-menopausal breast cancer survivors. . Cancer Res 2009;67(24):557S.
- [Background] Cheville AL, McGarvey CL, Petrek JA, Russo SA, Thiadens SR, Taylor ME. The grading of lymphedema in oncology clinical trials. Semin Radiat Oncol. 2003 Jul;13(3):214-25. doi: 10.1016/S1053-4296(03)00038-9. PMID 12903011
- [Background] Rogerino A, Grant LL, Wilcox H 3rd, Schmitz KH. Geographic recruitment of breast cancer survivors into community-based exercise interventions. Med Sci Sports Exerc. 2009 Jul;41(7):1413-20. doi: 10.1249/MSS.0b013e31819af871. PMID 19516160
- [Background] NLN Medical Advisory Commitee. Position Statement of the National Lymphedema Network. Topic: Lymphedema Risk Reduction Practices. In; 2005:1-2.
- [Background] Földi M, Földi, E., Strössenreuther, R.H.K., Kubik, S. Foldi's Textbook of Lymphology for Physicians and Lymphedema Therapists: For Physicians and Lymphedema Therapists. 2nd ed. Munich: Elsevier,Urban&FischerVerlag; 2006.
- [Background] Cornish BH, Thomas BJ, Ward LC. Effect of temperature and sweating on bioimpedance measurements. Appl Radiat Isot. 1998 May-Jun;49(5-6):475-6. doi: 10.1016/s0969-8043(97)00057-2. PMID 9569518
- [Background] Consensus Document on the Management of Cellulitis in Lymphoedema. British Lymphology Society and the Lymphedema Support Network, 2007. (Accessed October 26, 2009, at http://www.lymphoedema.org/lsn/consensus_on_cellulitis_dec_06.pdf.)
- [Background] Topic: Training of Lymphedema Therapists. National Lymphedema Network National Advisory Committee, 2005. (Accessed Access Date: September 17, 2008, 2008, at http://www.lymphnet.org/lymphedemaFAQs/positionPapers.htm.)
- [Background] Stanton AW, Northfield JW, Holroyd B, Mortimer PS, Levick JR. Validation of an optoelectronic limb volumeter (Perometer). Lymphology. 1997 Jun;30(2):77-97. PMID 9215977
- [Background] Tierney S, Aslam M, Rennie K, Grace P. Infrared optoelectronic volumetry, the ideal way to measure limb volume. Eur J Vasc Endovasc Surg. 1996 Nov;12(4):412-7. doi: 10.1016/s1078-5884(96)80005-0. PMID 8980428
- [Background] Labs KH, Tschoepl M, Gamba G, Aschwanden M, Jaeger KA. The reliability of leg circumference assessment: a comparison of spring tape measurements and optoelectronic volumetry. Vasc Med. 2000;5(2):69-74. doi: 10.1177/1358836X0000500202. PMID 10943582
- [Background] Coutts F, Grainger, A, Bulley, C. Perometer (400T) measurement of lower limb volume: Development of a standardised protocol. Physiotherapy 2007;93(Suppl 1):S670.
- [Background] Revill SI, Robinson JO, Rosen M, Hogg MI. The reliability of a linear analogue for evaluating pain. Anaesthesia. 1976 Nov;31(9):1191-8. doi: 10.1111/j.1365-2044.1976.tb11971.x. PMID 1015603
- [Background] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Norman SA, Miller LT, Erikson HB, Norman MF, McCorkle R. Development and validation of a telephone questionnaire to characterize lymphedema in women treated for breast cancer. Phys Ther. 2001 Jun;81(6):1192-205. PMID 11380275
- [Background] Fleck S, Kraemer W. Designing resistance training programs. 2nd ed. Champaign, IL: Human Kinetics; 1997.
- [Background] Bruce RA, Kusumi F, Hosmer D. Maximal oxygen intake and nomographic assessment of functional aerobic impairment in cardiovascular disease. Am Heart J. 1973 Apr;85(4):546-62. doi: 10.1016/0002-8703(73)90502-4. No abstract available. PMID 4632004
- [Background] Foster C, Jackson AS, Pollock ML, Taylor MM, Hare J, Sennett SM, Rod JL, Sarwar M, Schmidt DH. Generalized equations for predicting functional capacity from treadmill performance. Am Heart J. 1984 Jun;107(6):1229-34. doi: 10.1016/0002-8703(84)90282-5. No abstract available. PMID 6720550
- [Background] Hartwig JH, Bokoch GM, Carpenter CL, Janmey PA, Taylor LA, Toker A, Stossel TP. Thrombin receptor ligation and activated Rac uncap actin filament barbed ends through phosphoinositide synthesis in permeabilized human platelets. Cell. 1995 Aug 25;82(4):643-53. doi: 10.1016/0092-8674(95)90036-5. PMID 7664343
- [Background] Morales CR, Terry ES, Zackert WE, Montine TJ, Morrow JD. Improved assay for the quantification of the major urinary metabolite of the isoprostane 15-F(2t)-Isoprostane (8-iso-PGF(2alpha)) by a stable isotope dilution mass spectrometric assay. Clin Chim Acta. 2001 Dec;314(1-2):93-9. doi: 10.1016/s0009-8981(01)00637-4. PMID 11718683
- [Background] Subar AF, Midthune D, Kulldorff M, Brown CC, Thompson FE, Kipnis V, Schatzkin A. Evaluation of alternative approaches to assign nutrient values to food groups in food frequency questionnaires. Am J Epidemiol. 2000 Aug 1;152(3):279-86. doi: 10.1093/aje/152.3.279. PMID 10933275
- [Background] Subar AF, Thompson FE, Kipnis V, Midthune D, Hurwitz P, McNutt S, McIntosh A, Rosenfeld S. Comparative validation of the Block, Willett, and National Cancer Institute food frequency questionnaires : the Eating at America's Table Study. Am J Epidemiol. 2001 Dec 15;154(12):1089-99. doi: 10.1093/aje/154.12.1089. PMID 11744511
- [Background] Kriska AM, Knowler WC, LaPorte RE, Drash AL, Wing RR, Blair SN, Bennett PH, Kuller LH. Development of questionnaire to examine relationship of physical activity and diabetes in Pima Indians. Diabetes Care. 1990 Apr;13(4):401-11. doi: 10.2337/diacare.13.4.401. PMID 2318100
- [Background] Launois R, Mègnigbêto, A.C., Pocquet, K.,Alliot, F. A specific quality of life scale in upper limb lymphedema: the ULL-27 questionnaire. Lymphology 2002;35(Suppl):181-7.
- [Background] Hormes JM, Lytle LA, Gross CR, Ahmed RL, Troxel AB, Schmitz KH. The body image and relationships scale: development and validation of a measure of body image in female breast cancer survivors. J Clin Oncol. 2008 Mar 10;26(8):1269-74. doi: 10.1200/JCO.2007.14.2661. PMID 18323550
- [Background] Holm S. A simple sequentially rejective multiple test procedure. Scandinavian Journal of Statistics 1979;6:65-70.
- [Background] Hochberg Y. A sharper Bonferroni procedure for multiple tests of significance. Biometrika 1988;75:800-802.
- [Background] Singer J, Willett J. Applied Longitudinal Data Analysis. New York: Oxford University Press; 2003.
- [Background] Fitzmaurice G, Laird N, Ware J. Applied Longitudinal Analysis. Hoboken, New Jersey: Wiley; 2004.
- [Background] Troxel A. An index of local sensitivity to nonignorability. Statistica Sinica 2004;14:1221-37.
- [Background] Ma G, Troxel AB, Heitjan DF. An index of local sensitivity to nonignorable drop-out in longitudinal modelling. Stat Med. 2005 Jul 30;24(14):2129-50. doi: 10.1002/sim.2107. PMID 15909292
- [Background] Brewster AM, Hortobagyi GN, Broglio KR, Kau SW, Santa-Maria CA, Arun B, Buzdar AU, Booser DJ, Valero V, Bondy M, Esteva FJ. Residual risk of breast cancer recurrence 5 years after adjuvant therapy. J Natl Cancer Inst. 2008 Aug 20;100(16):1179-83. doi: 10.1093/jnci/djn233. Epub 2008 Aug 11. PMID 18695137
- [Background] Warren M, Schmitz KH. Safety of strength training in premenopausal women: musculoskeletal injuries from a two-year randomized trial. Am J Health Promot. 2009 May-Jun;23(5):309-14. doi: 10.4278/ajhp.07081584. PMID 19445432
- [Background] Powell KE, Heath GW, Kresnow MJ, Sacks JJ, Branche CM. Injury rates from walking, gardening, weightlifting, outdoor bicycling, and aerobics. Med Sci Sports Exerc. 1998 Aug;30(8):1246-9. doi: 10.1097/00005768-199808000-00010. PMID 9710864
- [Derived] Sturgeon KM, Brown JC, Sears DD, Sarwer DB, Schmitz KH. WISER Survivor Trial: Combined Effect of Exercise and Weight Loss Interventions on Inflammation in Breast Cancer Survivors. Med Sci Sports Exerc. 2023 Feb 1;55(2):209-215. doi: 10.1249/MSS.0000000000003050. Epub 2022 Sep 29. PMID 36170550
- [Derived] Schmitz KH, Troxel AB, Dean LT, DeMichele A, Brown JC, Sturgeon K, Zhang Z, Evangelisti M, Spinelli B, Kallan MJ, Denlinger C, Cheville A, Winkels RM, Chodosh L, Sarwer DB. Effect of Home-Based Exercise and Weight Loss Programs on Breast Cancer-Related Lymphedema Outcomes Among Overweight Breast Cancer Survivors: The WISER Survivor Randomized Clinical Trial. JAMA Oncol. 2019 Nov 1;5(11):1605-1613. doi: 10.1001/jamaoncol.2019.2109. PMID 31415063
- [Derived] Winkels RM, Sturgeon KM, Kallan MJ, Dean LT, Zhang Z, Evangelisti M, Brown JC, Sarwer DB, Troxel AB, Denlinger C, Laudermilk M, Fornash A, DeMichele A, Chodosh LA, Schmitz KH. The women in steady exercise research (WISER) survivor trial: The innovative transdisciplinary design of a randomized controlled trial of exercise and weight-loss interventions among breast cancer survivors with lymphedema. Contemp Clin Trials. 2017 Oct;61:63-72. doi: 10.1016/j.cct.2017.07.017. Epub 2017 Jul 21. PMID 28739540
- [Derived] Dean LT, Kumar A, Kim T, Herling M, Brown JC, Zhang Z, Evangelisti M, Hackley R, Kim J, Cheville A, Troxel AB, Schwartz JS, Schmitz KH. Race or Resource? BMI, Race, and Other Social Factors as Risk Factors for Interlimb Differences among Overweight Breast Cancer Survivors with Lymphedema. J Obes. 2016;2016:8241710. doi: 10.1155/2016/8241710. Epub 2016 Jun 28. PMID 27433356